CLINICAL TRIAL: NCT07082647
Title: The Importance of Different Types of Feedback in Sports Pedagogy
Brief Title: Different Types of Feedback in Sports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Vesile Şahiner Güler, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERU-SAGENS-VSG-02
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Training Effectiveness; Motor Skills Development; Motor Learning
Keywords: Learning; Motor Learning; Motor Skill; Feedback

STUDY DESIGN:
Intervention Model Description: Interventional Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mixed Group (Experimental): Group 1 (Mixed Feedback Group n=20) is the group in which both verbal and visual (video-supported) feedback methods were used together while applying the training program to the gymnasts.
  Interventions: Behavioral: Mixed feedback method
- Visual Feedback Group (Experimental): Group 2 is the group where the gymnasts are provided with visual feedback in some way throughout the training program. (Visual Feedback Group = 20)
  Interventions: Behavioral: Visual feedback method
- Verbal Group (Experimental): Group 3 (Verbal Group n=20) is the group in which verbal feedback methods are predominantly used when applying the training program to gymnasts.
  Interventions: Behavioral: Verbal feedback method

INTERVENTIONS:
Behavioral: Mixed feedback method — Feedback (technical correction) method in which both visual and verbal feedback are predominantly used in the feedback given to the participants throughout the training program.
  Arms: Mixed Group
Behavioral: Visual feedback method — Feedback (technical correction) method in which visual feedback is predominantly used in the feedback given to gymnasts throughout the training program.
  Arms: Visual Feedback Group
Behavioral: Verbal feedback method — Feedback (technical correction) method in which verbal feedback is predominantly used in the feedback given to gymnasts throughout the training program.
  Arms: Verbal Group

SUMMARY:
The aim of the study is to examine the effects of mixed (visual + verbal) feedback, visual feedback and verbal feedback methods applied to gymnasts between the ages of 7-11 on the front scale, back scale (knee-knee), back scale (shoulder-knee) and split jump elements by kinematic methods.

DETAILED DESCRIPTION:
The participants were asked to perform the measured movements one by one during the training, and feedback was given to each participant one by one. In the study, kinematic analyzes were made by taking video recordings (measurements taken at 3 different times) of the elements performed by the participants in gymnastics. As a result, it was determined that the most effective feedback method for all elements except the split jump element was the mixed method, the most effective method for the split jump was the visual method, and the least effective method for all elements was the verbal method.The students were given the following training program (2 days a week) for 8 weeks and each group was given the same training curriculum with its own feedback method; Weeks: 1 Lesson 1:Running, Animal Walks, Forward Roll, Front Scale, Back Scale, Split Jump, Bridge, Middle Split, Front Splits Lesson 2: Running, Animal Walks, Forward Roll, Backward Roll, Front Scale, Back Scale, Split Jump, Balance (static) Exercises, Bridge, Middle Split, Front Splits Weeks:2 Lesson 1: Running, Animal Walks, Forward Roll, Backward Roll, Front Scale, Back Scale, Split Jump, Static Strength Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Animal Walks, Roll Exercises, Cartwheel, Front Scale, Back Scale, Split Jump, Staircase Exercise, Bridge, Middle Split, Front Splits

Weeks 3:

Lesson 1: Running, Stretching Exercises, Animal Walks, Roll Exercises, Cartwheel, Front Scale, Back Scale, Split Jump, Plyometric Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Animal Walks, Cartwheel, Front Scale, Back Scale, Split Jump, Balance (static) Exercise, Bridge, Middle Split, Front Splits Weeks:4 Lesson 1: Scale, Back Scale, Split Jump, Dynamic Strength Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Animal Walks, Cartwheel, Handstand Exercise, Front Scale, Back Scale, Split Jump, Stretching Exercise, Bridge, Middle Split, Front Splits Weeks:5 Lesson 1: Running, Stretching, Animal Walks, Roll Exercises, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Static Strength Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Stretching, Animal Walks, Roll Exercises, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Staircase Exercises, Bridge, Middle Split, Front Splits Weeks:6 Lesson 1:Running, Stretching, Animal Walks, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Plyometric Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Animal Walks, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Bridge, Middle Split, Front Splits Weeks: 7 Lesson 1: Running, Stretching, Animal Walks, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Dynamic Strength Exercises, Bridge, Middle Split, Front Splits Lesson 2: Stretching, Animal Walks, Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Running Exercise, Bridge, Middle Split, Front Splits Weeks:8 Lesson 1: Cartwheel, Handstand, Front Scale, Back Scale, Split Jump, Static Strength Exercises, Bridge, Middle Split, Front Splits Lesson 2: Running, Stretching, Animal Walks, An overview, Back Scale, Split Jump, Bridge, Middle Split, Front Splits.

As a result of the training program, the development of the gymnasts' Front Scale, Back Scale (Knee-Knee), Back Scale (Shoulder-Knee) and Split jump movements was examined.

Body weight measurement The participants' body weights were measured with a Xiaomi electronic scale with an accuracy of ±0.1 kg Participants' BMI was calculated as body mass (kg)/height (m2).

Height measurement Participants' heights and leg lengths measurements were measured using a Fisco brand meter ±0.1 (cm)

ELEMENTS AND ANALYSIS Front scale The basic posture begins with position and posture. With the arms up and one foot stretched above 90 degrees, the other foot at the bottom rises up to the toes and waits steadily for two seconds Back scale The movement begins with a standing position and a basic posture. In gymnastics, it is a posture in which one of the feet is on the ground and the body weight is on one leg. In the scale pose, the other leg is expected to lift up tautly. The arms are open at the sides and shoulder level. The body and arms are parallel to the ground Split jump The split jump movement, the arms are positioned above, and the legs are opened forward and back, creating a 180-degree angle KINOVEA VIDEO ANALYSING The video recordings of the athletes during the lessons were analyzed with the Kinovea program: Kinovea is a free software application that analyzes, compares, and evaluates movement. It is often used to evaluate an athlete's progress in training For kinematic analysis, recordings were made with a Redmi Note 11 mobile phone, and a Lenovo G5 laptop was used for the relevant analysis.

Front scale analysis The highest angular distance between the knee joints and the two legs was measured on the front scale (stance over 90 degrees with the leg forward).

Back scale analysis (knee-knee) and (shoulder-knee) The angle between the hind leg knee joint (knee-knee) and the shoulder and the highest angular (shoulder-knee) distance between the two legs were recorded in the scale movement. Although the back scale (knee-knee) and back scale (shoulder-knee) elements were tested on the same movement, their angular values were recorded and evaluated independently.

Split jump analysis When the jump occurred in the split jump movement, the highest angle that could be reached between the two legs and the angles of the knee joints in the relevant position were recorded.

ANALYSIS OF DATA The data used in the research were analyzed through the SPSS 27 program. The normality distributions of the data obtained with the Shapiro Wilk test are examined. Since the data obtained showed a parametric distribution, a one-way analysis of variance was applied for comparison between groups. For intragroup comparisons, analysis of variance was used for repeated measurements, and the Bonferroni test was used to reveal the source of the difference.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7-11 years old
* Being a female
* Being an active gymnast

Exclusion Criteria:

* Being outside between the ages of 7-11
* Being a man
* Not being involved in gymnastics

Ages: 7 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — It was appropriate for female gymnasts to participate in the study.
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of feedback methods. | Measurements were taken three times: before the training program was implemented, at the end of the 4th week of the training program, and at the end of the 8th week after the training program was completed.
  All feedback methods (each group having its own method) were applied to athletes who received the same gymnastics training 2 days a week for 8 weeks, in addition to their training. The unit of all measurements is the angle degree. This refers to the measurement of the angle between the designated points (knee, shoulder) when the relevant gymnastic element is performed. ELEMENTS AND ANALYSIS Front scale The basic posture begins with position and posture. With the arms up and one foot stretched above 90 degrees, the other foot at the bottom rises up to the toes and waits steadily for two seconds Back scale The movement begins with a standing position and a basic posture. In gymnastics, it is a posture in which one of the feet is on the ground and the body weight is on one leg. In the scale pose, the other leg is expected to lift up tautly. The arms are open at the sides and shoulder level. The body and arms are parallel to the ground Split jump The split jump movement, the arms are pos

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Behzat Turan, Associate Professor, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Talas, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No